CLINICAL TRIAL: NCT02387606
Title: A Phase 2a, Randomized, Double-blinded, Placebo-Controlled Study to Evaluate the Antiviral Activity, Safety, and Pharmacokinetics of Repeated Doses of Orally Administered JNJ 53718678 Against Respiratory Syncytial Virus Infection in the Virus Challenge Model in Healthy Adult Subjects
Brief Title: Study to Evaluate Antiviral Activity, Safety, and Pharmacokinetics of Repeated Doses of Orally Administered JNJ 53718678 Against Respiratory Syncytial Virus Infection.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106786; 2014-005041-41 (EudraCT Number); 53718678RSV2001 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Infections; Placebo; Antiviral activity; JNJ-53718678
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive placebo or JNJ-53718678 500 milligram (mg) or 200 mg once daily for 7 days.
  Interventions: Drug: Placebo; Drug: JNJ-53718678
- Cohort 2 (Experimental): Participants will receive placebo or JNJ-53718678; dosing regimen in Cohort 2 will be decided based on Cohort 1 results.
  Interventions: Drug: Placebo; Drug: JNJ-53718678
- Cohort 3 (Experimental): Participants will receive placebo or JNJ-53718678, 75 mg once daily for 7 days.
  Interventions: Drug: Placebo; Drug: JNJ-53718678

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo once daily.
Drug: JNJ-53718678 — Participants will receive JNJ-53718678 as 20 milliliter (mL) (200 mg) or 50 mL (500 mg) oral solution (containing 10 mg JNJ-53718678 per mL) in Cohort 1. JNJ-53718678 dose in Cohort 2 will be decided based on Cohort 1 results. JNJ-53718678 as 7.5 mL (75 mg) oral solution (containing 10 mg JNJ-53718678 per mL) in Cohort 3.

SUMMARY:
The purpose of this study is to evaluate the antiviral effect of repeated oral dosing of JNJ 53718678 compared to placebo in healthy adult participants infected through inoculation with respiratory syncytial virus (RSV)-A Memphis 37b virus.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo-controlled, single-center study of JNJ 53718678 in healthy adult participants. Study consists of 3 phases: Screening (Day -56 and Study Day -3 prior to the planned date of virus inoculation/challenge on Study Day 0), quarantine (includes challenge on Day -1 or -2 and treatment for 7 days), and follow-up (Day 15 and 28). Participants will be admitted to the quarantine unit on Study Day -1 or - 2 and will be inoculated (intranasal) with the RSV-A Memphis 37b virus on Study Day 0. Participants will be evaluated in 3 cohorts: Cohort 1 and Cohort 3 (participants will be dosed with JNJ-53718678 or placebo for 7 days) and Cohort 2 (for up to 7 days [Dosing Days 1-x] [x will be determined based on the results from Cohort 1]). Participants will be randomized and JNJ-53718678/placebo dosing will be started after RSV presence in nasal wash has been detected by polymerase chain reaction (PCR). After completion of Cohort 1, data will be reviewed (unblinded) and the antiviral activity, safety, pharmacokinetic, clinical symptom and mucus weight data will be evaluated, based on which Cohort 2 will be initiated. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must be of non-childbearing potential: postmenopausal for at least 2 years or surgically sterile or otherwise incapable of becoming pregnant
* Female participants, except for postmenopausal women, must have a negative serum pregnancy test at screening
* Participants must agree to comply with contraceptive measures as mentioned in protocol
* Participants must be sero-suitable for respiratory syncytial virus (RSV) within 57 days prior to inoculation
* Participants must be non-smokers for at least one month prior to screening and participants must have a negative cotinine test at screening

Exclusion Criteria:

* Participants with a past history of heart arrhythmias (extrasystoli, tachycardia at rest) or of risk factors for Torsade de Pointes syndrome
* Participants with a history or evidence of abuse of alcohol, barbiturates, amphetamines, recreational or narcotic drug use within the past 3 months, which in the Investigator's opinion would compromise participant's safety and/or compliance with the study procedures
* Participants with current human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection at screening
* Participants with current hepatitis A infection, or hepatitis B virus (HBV) infection, or hepatitis C virus (HCV) infection (confirmed by HCV antibody) at screening
* Participants with active acute respiratory infection at admission (Study Day -1 or -2)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2015-09-21 (Actual); Study Completion 2015-10-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Viral Load-time Curve (VL AUC) | up to Follow-up (Day 28)
  VL AUC for RSV-A Memphis 37b will be determined by quantitative reverse transcriptase -polymerase chain reaction (qRT-PCR) assay of nasal wash. The VL AUC will be calculated based on the viral load values measured 2 times per day, starting with the last value prior to first dosing, and ending with the last available value before discharge.

SECONDARY OUTCOMES:
Area Under the Viral Load-time Curve (VL AUC) Determined by Plaque Forming Unit (PFU) Assay | Baseline up to Follow-up (Day 28)
  VL AUC for RSV-A Memphis 37b will be determined by PFU assay of nasal wash.
Viral Load Over Time | Baseline up to Follow-up (Day 28)
Peak Viral Load | Baseline up to Follow-up (Day 28)
Time To Peak Viral Load | Baseline up to Follow-up (Day 28)
  Time to peak viral load will be reported.
Area Under the Viral Load-time Curve (VL AUC) From Time 0 to 24 Hours after First Dose | 24 hours after first dose
Area Under the Viral Load-time Curve (VL AUC) From Time 0 to 48 Hours after First Dose | 48 hours after first dose
Time to Non-detectability of Virus | Baseline up to Follow-up (Day 28)
  Time to non-detectability of virus from first administration of study drug will be assessed.
Total Clinical Symptom Score | Admission (Day -1 or -2) up to Day 13
  Total clinical symptom score will be assessed using a composite of 10 self-reported symptoms on the Symptom Diary Card. The Investigator will review the participant's SDC entries on a daily basis after the administration of challenge virus inoculum. Total Clinical Symptom Score ranges from 0 (no symptoms) to 3 (not well).
Time to Peak Symptom Score After Viral Inoculation | Admission (Day -1 or -2) up to Day 13
Mucus Weight | Baseline up to Day 13
Tissue Count | Baseline up to Day 13
Sequence Analysis of the Rsv-A Memphis 37b Genome | Baseline and post-Baseline
Forced Expiratory Volume in 1 Second (FEV1) Measured by Spirometry | Baseline up to Follow-up (Day 28)
  FEV1 is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.
Forced Vital Capacity (FVC) Measured by Spirometry | Baseline up to Follow-up (Day 28)
  FVC is the total volume of air expired after a full inspiration.
FEV1/FVC Ratio | Baseline up to Follow-up (Day 28)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- London, United Kingdom

REFERENCES:
- [Derived] Stevens M, Rusch S, DeVincenzo J, Kim YI, Harrison L, Meals EA, Boyers A, Fok-Seang J, Huntjens D, Lounis N, Mari N K, Remmerie B, Roymans D, Koul A, Verloes R. Antiviral Activity of Oral JNJ-53718678 in Healthy Adult Volunteers Challenged With Respiratory Syncytial Virus: A Placebo-Controlled Study. J Infect Dis. 2018 Jul 24;218(5):748-756. doi: 10.1093/infdis/jiy227. PMID 29684148